CLINICAL TRIAL: NCT06967064
Title: The Application of Lidocaine Cream on Oral Secretions of LMA Removal During the Recovery Period in Ophthalmic Surgical Patients Under General Anesthesia: a Randomized Controlled Trial
Brief Title: The Application of Lidocaine Cream on Oral Secretions of LMA Removal During the Recovery Period in Ophthalmic Surgical Patients Under General Anesthesia
Acronym: LICOS
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: The study was proactively suspended to ensure alignment with all applicable regulatory filing procedures. This decision was made to maintain adherence to institutional and compliance standards prior to study initiation.
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Zhu Yanling, Attending doctor of anesthesiology, Zhongshan Ophthalmic Center, Sun Yat-sen University, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2000035364
Record Dates: First submitted 2025-04-22; First posted 2025-05-13 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Airway Complication of Anaesthesia; Laryngeal Mask Airway Removal; Anesthesia Emergence; Secretion; Excess, Salivation; Ophthalmic Surgery; General Anesthesia
Keywords: airway complication; oral secretions; laryngeal mask airway; general anesthesia; ophthalmic surgery
MeSH Terms: conditions — Sialorrhea

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- The uniform application group (group U) (Experimental): 1 ml of lidocaine cream will be evenly applied to the posterior surface of the LMA cuff before insertion
  Interventions: Drug: lidocaine cream
- The non-uniform application group (group N) (Experimental): 1 mL of lidocaine cream will be applied to the posterior surface without ensuring uniform coverage before insertion
  Interventions: Drug: lidocaine cream
- The control group (group C) (Sham Comparator): No lidocaine cream will be applied to the LMA
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: lidocaine cream — Group U receives 1 mL of lidocaine cream extracted using a syringe and evenly applied across the entire posterior surface of the LMA cuff by carefully spreading the cream to ensure uniform coverage, while Group N receives 1 mL of lidocaine cream also extracted using a syringe but applied without ensuring even distribution, resulting in a patchy or non-uniform application.
  Arms: The non-uniform application group (group N); The uniform application group (group U)
Other: Placebo — No lidocaine cream will be applied to the LMA
  Arms: The control group (group C)

SUMMARY:
The application of lidocaine cream on oral secretions of LMA removal during the recovery period in ophthalmic surgical patients under general anesthesia: a randomized controlled trial

DETAILED DESCRIPTION:
During the recovery from general anesthesia, patients commonly experience heightened oral secretions, which can elevate intraocular pressure (IOP) due to coughing and potentially lead to the infiltration of secretions into the surgical site via the nasolacrimal duct, increasing the risk of endophthalmitis. This study is aimed to investigate whether applying lidocaine cream to the laryngeal mask airway (LMA) reduces oral secretions during emergence from general anesthesia in ophthalmic surgery patients.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 to 60 years;
* With American Society of Anesthesiologists (ASA) physical status I or II;
* Scheduled to undergo ophthalmic surgery following general anesthesia with LMA.

Exclusion Criteria:

* Contraindications to LMA use;
* A history of upper respiratory tract infection within one week prior to surgery;
* Persistent pharyngeal symptoms (eg. throat irritation, dryness, or chronic cough, etc.) lasting ≥ 3 months;
* Severe gastroesophageal reflux disease;
* Morbid obesity, defined as a body mass index ≥ 40 kg/m2;
* A predicted difficult airway (eg. a history of difficult airway, mouth opening < 3 cm, Mallampati class 4, limited neck extension or cervical spine disease);
* Presence of structural abnormalities, masses, infections, or scarring in the oral cavity or oropharynx;
* Known contraindications to lidocaine cream;
* Two or more failed attempts at LMA insertion;
* Intraoperative administration of anticholinergic agents;
* Any other condition present likely to influence the study outcomes.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2025-05-15 (Actual); Primary Completion 2025-05-22 (Actual); Study Completion 2025-05-22 (Actual)

PRIMARY OUTCOMES:
The volume of oral secretions | Assessed during the phase of anesthesia emergence, from the discontinuation of anesthetic agents to eye opening or purposeful movement; and reported up to 4 weeks.
  Oral secretions will be collected during the phase of anesthesia emergence. In the PACU, oral and nasopharyngeal secretions are gently suctioned using a negative pressure aspirator during the phase of emergence. Subsequently, 50 ml of normal saline is used to flush the suction tubing. The volume of oral secretions (ml) is calculated as the total volume in the suction canister minus 50 ml.

SECONDARY OUTCOMES:
The time completion of LMA insertion | Assessed from holding the airway tube to successful insertion of the LMA; and reported up to 4 weeks.
Oropharyngeal leak pressure (OLP) | Assessed after the completion of LMA insertion; and reported up to 4 weeks.
  OLP is measured by setting the expiratory valve to 30 cmH2O at a gas flow rate of 3 L/min, recording the maximum inflation pressure when a noise of gas leakage is heard in the oropharynx via a stethoscope
Time to LMA removal | Assessed from discontinuation of anesthetic agents to LMA removal; and reported up to 4 weeks.
Time to emergence | Assessed from the discontinuation of anesthetic agents to eye opening or purposeful movement; and reported up to 4 weeks.
PACU recovery time | Assessed from arrival in the PACU until the modified Aldrete score achieved at least 9; and reported up to 4 weeks.
Postoperative airway complications | Assessed at the time of LMA removal; and reported up to 4 weeks.
  Postoperative airway complications, including coughing, laryngospasm, or blood on device, will be recorded at the time of LMA removal
Pharyngeal complications | Assessed at 1 h and 24 h postoperatively; and reported up to 4 weeks.
  Pharyngeal complications, such as sore throat, dysphagia, or hoarseness, will be collected
The level of sore throat | Assessed at 1 h and 24 h postoperatively; and reported up to 4 weeks.
  The level of sore throat will be graded as follows: none, no sore throat; mild, pain with deglutition; moderate, pain constantly present and increasing with deglutition; severe, pain interfering with eating and requiring analgesic medication
Ocular and other complications | Assessed within 48 h after the surgery; and reported up to 4 weeks.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Seo JH, Cho CW, Hong DM, Jeon Y, Bahk JH. The effects of thermal softening of double-lumen endobronchial tubes on postoperative sore throat, hoarseness and vocal cord injuries: a prospective double-blind randomized trial. Br J Anaesth. 2016 Feb;116(2):282-8. doi: 10.1093/bja/aev414. PMID 26787799
- [Background] van Esch BF, Stegeman I, Smit AL. Comparison of laryngeal mask airway vs tracheal intubation: a systematic review on airway complications. J Clin Anesth. 2017 Feb;36:142-150. doi: 10.1016/j.jclinane.2016.10.004. Epub 2016 Dec 3. PMID 28183554
- [Background] Zhu Y, Shen W, Lin Y, Huang T, Xie L, Yang Y, Chen H, Gan X. Cricoid-mental distance-based versus weight-based criteria for size selection of classic laryngeal mask airway in adults: a randomized controlled study. J Clin Monit Comput. 2019 Oct;33(5):759-765. doi: 10.1007/s10877-019-00308-w. Epub 2019 Apr 8. PMID 30963460
- [Background] Park JJ, Huh H, Yoon SZ, Lim HJ, Go DY, Cho JE, Lee J, Park J, Kim HC. Two-handed jaw thrust decreases postoperative sore throat in patients undergoing double-lumen endobronchial intubation: A randomised study. Eur J Anaesthesiol. 2020 Feb;37(2):105-112. doi: 10.1097/EJA.0000000000001149. PMID 31860598
- [Background] Zhu YL, Shen WH, Chen QR, Ye HJ, Huang JX, Kang Y, Chi W, Gan XL. Desflurane anesthesia compared with total intravenous anesthesia on anesthesia-controlled operating room time in ambulatory surgery following strabotomy: a randomized controlled study. Chin Med J (Engl). 2020 Apr 5;133(7):779-785. doi: 10.1097/CM9.0000000000000728. PMID 32149764